CLINICAL TRIAL: NCT03445962
Title: SLEEP APNEA SYNDROME AND TRISOMY 21 : Exploration of the Predictive Factors in the Population With Trisomy 21
Brief Title: 19/5000 (SYNAPSOT21) Predictive Factors of Sleep Apnea Syndrome in Down Syndrome
Acronym: SYNAPSOT21
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.161
Record Dates: First submitted 2018-01-17; First posted 2018-02-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Down Syndrome; Sleep Apnea, Obstructive; Polysomnography
Keywords: Autonomic nervous system; Heart rate variability; Physical Activity; exercise; biological parameters; cephalometry; body composition; actigraphy; motor capacity; physical fitness; aerobic capacity; seismocardiography
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Down Syndrome (DS): Assessment of OSAS predictive factors in Down Syndrome without or without OSAS
  Interventions: Diagnostic Test: Assessment of OSAS predictive factors

INTERVENTIONS:
Diagnostic Test: Assessment of OSAS predictive factors — All subjects of the two groups realized the same assessment:
  * Anthropometric evaluation
  * biological examination (hormonal, inflammatory and complete blood count, and lipidic profile)
  * rest electrocardiogram
  * motor assessment (strenght, flexibility and balance)
  * actigraphy
  * Autonomic nervous system assessment during sleep
  * Autonomic nervous system assessment during head up tilt test before and after physical exercise
  * maximal treadmill test (VO2 max measure)
  * polysomnography
  * seismocardiography
  * questionnaires :sleep and physical activity

SUMMARY:
The obstructive sleep apnea syndrome (OSAS) is frequently reported in subjects with trisomy 21. The consequences of this syndrome are expressed in various disorders such as cognitive and cardiovascular alterations. It is also reported a premature exhaustion with the achievement of various professional or recreational activities, as well as an increase in the frequency of daytime sleepiness. In trisomy 21, there are factors that are systematically associated with obstructive apnea. The identification of these factors would make it possible to diagnose OSAS earlier, under-diagnosed in the population with trisomy 21 even though these OSAS are associated with increased cardiovascular risks.

The aim of this study is to identify the predictive factors associated with sleep apnea in the trisomy population in order to propose early detection.

OSAS treatment in a young adult with Down syndrome could reduce physical fatigue apparition during various activities, reduce daytime sleepiness, and have a positive impact on physical fitness, and therefore more broadly on health.

DETAILED DESCRIPTION:
The predictive factors for OSA that will be studied are: physical activity level, dentofacial disharmonies, blood parameters, motor disabilities, heart rate variability parameters measured during sleep and during autonomic nervous stimulation by orthostatic test.

All these factors will be linked to the data obtained by:

1. polysomnography
2. by the joint use of seismocardiography

OSAS lead to many associated disorders, which identified early can be better supported to limit the deleterious effects of this OSAS:

(i) a sudden and repeated activation of the sympathetic nervous system triggered by sleep fragmentation (ii) intermittent hypoxia associated with OSAS may increase insulin resistance through the involvement of an inflammatory state and oxidative stress.

(iii) a significant level of diurnal fatigue limiting activities, thus promoting a sedentary lifestyle and increasing cardiovascular risk factors.

Several secondary objectives will therefore be studied:

1. Can OSAS be predicted by the existence of autonomic dysfunction?
2. Can OSAS be predicted by specific biological disturbances?
3. Can OSAS be predicted by the presence of a specific cranial structure?
4. Can OSAS be predicted by an insufficient level of physical activity?

Finally does the use seismocardiography make it possible to identify quickly and early these risk factors linked to OSAS?

ELIGIBILITY:
Inclusion Criteria:

Subjects with Down syndrome, able to practice physical activity all participants have received information all have signed the consent form

Exclusion Criteria:

* pregnant women
* Pharmacological treatment altering autonomic nervous system (ANS)
* Contra-indication to physical exercise, such as atlanto-axial instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Down syndome voluntary to participated
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Identification of predictive factors associated to obstructive sleep apnea syndrome in DS subjects | 4 months
  OSAS will be diagnosed with polysomnography and seismocardiography. AHI threshold will be 15 to diagnose an OSAS (score).

SECONDARY OUTCOMES:
dysautonomia role on OSAS in DS | 1 day
  Cardiac response during exercise (existence of chronotropic incompetence
  %HR(reserve)lower than 80%)
Investigation of autonomic nervous system | 1 day
  spectral variations of blood pressure and heart rate variability during head-up tilt test : (spectral density in ms² and normalized units)
Oxygenation and dysautonomia | 1 day
  Cerebral and peripheral oxygenation parameters measured with near-infrared spectroscopy during head-up tilt test (delta Hbtot between supine and head up tilt positions)
  - Cardiac response during exercise (existence of chronotropic incompetence)
Investigation of dysautonomia during sleep | 3 nignts
  spectral variations of heart rate variability (spectral density in ms² and normalized units)
Biological profile | 1 day
  Disorders in blood parameters will be assessed by different inflammatory, corticotropic, thyroid and glycemic values in comparison with reference values.
anthropometric characteristics role on OSAS in DS | 1 day
  Existence of morphologic specificities will be investigated:
  Craniofacial abnormalities with orthopantomogram (degree)
Metabolic syndrome | 1 day
  Existence of morphologic specificities will be investigated:
  Neck, waist and hips circumferences (cm)
morphologic parameters | 1 day
  Existence of morphologic specificities will be investigated:
  Body fat composition (%)
Quantification of physical activity | 15 days
  Physical activity level will be assessed with actigraphy (min or h per day)
Motor skills | 15 days
  motor capacities : strength (explosive leg power (cm) and handgrip measure), flexibility (cm), balance (cm)
questionnaire of physical activity | 15 days
  G- PAQ and parental perceptions of physical activity (score)
Sleep questionnaire | 15 days
  Epworth and Pittsburg questionnaire (score)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DOUTRELEAU, MD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Échirolles, France

REFERENCES:
- [Background] Leti T, Guinot M, Favre-Juvin A, Bricout VA. Difference of catecholamine responses to exercise in men with trisomy 21, with or without chronotropic incompetence. Physiol Behav. 2015 Apr 1;142:97-103. doi: 10.1016/j.physbeh.2015.02.007. Epub 2015 Feb 4. PMID 25660758
- [Background] Bricout VA, Guinot M, Faure P, Flore P, Eberhard Y, Garnier P, Juvin AF. Are hormonal responses to exercise in young men with Down's syndrome related to reduced endurance performance? J Neuroendocrinol. 2008 May;20(5):558-65. doi: 10.1111/j.1365-2826.2008.01695.x. Epub 2008 Mar 15. PMID 18363810
- [Background] Flore P, Bricout VA, van Biesen D, Guinot M, Laporte F, Pepin JL, Eberhard Y, Favre-Juvin A, Wuyam B, van de Vliet P, Faure P. Oxidative stress and metabolism at rest and during exercise in persons with Down syndrome. Eur J Cardiovasc Prev Rehabil. 2008 Feb;15(1):35-42. doi: 10.1097/HJR.0b013e3282f2bff3. PMID 18277183
- [Result] Nguyen TD, Baillieul S, Guinot M, Doutreleau S, Bricout VA. Classification of Factors Effect on Sleep in Individuals with Down Syndrome. Brain Sci. 2021 Nov 12;11(11):1500. doi: 10.3390/brainsci11111500. PMID 34827499